CLINICAL TRIAL: NCT01563003
Title: Cognitive Behavioral Therapy for Anxiety Disorders in Adolescents With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AASD-2012
Record Dates: First submitted 2012-03-22; First posted 2012-03-26 (Estimated); Results first posted 2015-04-17 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Autism; Asperger's Syndrome; Pervasive Developmental Disorder Not Otherwise Specified; Generalized Anxiety Disorder; Social Phobia; Separation Anxiety Disorder; Obsessive-compulsive Disorder
Keywords: Autism; Asperger's Syndrome; Pervasive Developmental Disorder Not Otherwise Specified; Treatment; Cognitive-behavioral therapy; Anxiety; Children; Therapy
MeSH Terms: conditions — Autistic Disorder; Asperger Syndrome; Generalized Anxiety Disorder; Phobia, Social; Anxiety, Separation; Obsessive-Compulsive Disorder; Anxiety Disorders | interventions — Cognitive Behavioral Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavioral Therapy Condition (Experimental): This arm is the experimental condition; it consists of 16 weekly CBT sessions. This intervention program is flexible in nature and employs a modular format. Despite the added flexibility of the modular format, a minimum of three sessions are spent on basic coping skills and eight are spent on in vivo exposures to ensure an adequate and comparable dose of the core elements of CBT for anxiety across cases
  Interventions: Other: Cognitive Behavioral Therapy
- Treatment as Usual (Active Comparator): This arm acts as the comparison condition. Participants randomized to this arm will be instructed to continue receiving their prior interventions as recommended by their providers (e.g., psychotherapy, social skills training, behavioral interventions, family participation in family therapy or a parenting class, or pharmacological interventions). Treatment changes (e.g., medication increase, starting psychotherapy in the community) are not prohibited and will be monitored. Thus, treatment will continue as it would in standard practice; and will be monitored through periodic study assessment.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: Cognitive Behavioral Therapy — This condition involves 16 weekly CBT sessions.
  Arms: Cognitive Behavioral Therapy Condition
Other: Treatment as usual — This condition allows participants to seek out various services. Considering the number of possible treatment options, there is no way to identify or list them.
  Arms: Treatment as Usual

SUMMARY:
Due to the considerable prevalence of anxiety in youth with autism spectrum disorders, this study seeks to establish the efficacy of a modified cognitive behavioral therapy protocol in 50 adolescents versus other available treatment options.

DETAILED DESCRIPTION:
This study will further examine a treatment plan for adolescents with autism spectrum disorderS (ASD) and anxiety. Many children who have an autism spectrum disorder experience substantial anxiety that can cause impairment above that of an ASD alone. Few studies have examined effective treatment options for anxiety in this population. In typically developing youth, Cognitive Behavioral Therapy (CBT) is considered the gold standard for treating anxiety. But, in order to address the unique needs of children with ASD, this study utilizes a modified CBT treatment plan which includes social skills and parent training. In our past studies, this cognitive-behavioral treatment plan has been effective in kids with ASD and anxiety compared to kids who did not receive any treatment.The current study compares this modified treatment plan to other treatment options in the community. The experimental component of this study is being assigned to 1 of 2 groups. The first group will receive CBT immediately for a period of 16 weeks. The second group will have to wait 16 weeks before receiving CBT. During this time period, children may receive any other services in the community. Overall, all adolescents receive the same type of therapy; it's matter of whether he/she receives it immediately or after a wait period. Sixteen weekly sessions comprise CBT. All therapy and assessments associated with this study will be free of charge.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient children with an autism spectrum disorder (see #2 below) between the ages 11-16 years.
2. Meets criteria for a diagnosis of autism, Asperger syndrome (AS), or PDD-NOS using scores from the Autism Diagnostic Interview-Revised and the Childhood Autism Rating Scale.
3. Meets DSM-IV criteria for a diagnosis of one of the following anxiety disorders: separation anxiety disorder (SAD), generalized anxiety disorder (GAD), social phobia, or obsessive compulsive disorder (OCD) as determined by the ADIS-IV-C/P (with CSR 4) and all available information.
4. Minimum score of 13 on the PARS Severity Scale; this score indicates clinically significant anxiety symptom severity (RUPP, 2002) and has been used in recent major clinical trials (e.g., Walkup et al., 2008).
5. Child has a Full Scale and Verbal Comprehension IQ > 80 as assessed on a commonly used IQ test.
6. Subjects with co-morbid depression, ADHD, tic disorder or disruptive behavior disorders will be acceptable as long as the anxiety disorder is primary (i.e., most impairing/distressing).

Exclusion Criteria:

1. Receiving concurrent psychotherapy, social skills training, or behavioral interventions (e.g., applied behavior analysis). Families will have the option of discontinuing such services to enroll in the study.
2. New Treatments: Initiation of an antidepressant within 12 weeks before study enrollment or an antipsychotic 6 weeks before study enrollment. No new alternative medications, nutritionals or therapeutic diets within 6 weeks of study enrollment.
3. Established Treatment changes: Any change in established psychotropic medication (e.g., antidepressants, anxiolytics) within 8 weeks before study enrollment (6 weeks for antipsychotic). Alternative medications that might have behavioral effects must be stable for 6 weeks prior to the study baseline assessment. Any medications that the adolescent is on must remain stable during treatment. If a potential participant is taking psychotropic medication at the time of the phone evaluation or the first in-person study assessment and wishes to discontinue this medication to enter the study, the patient will be asked to discuss this option with their prescribing physician to determine whether medication discontinuation would be safe and in the adolescent's best interest. In addition, we will obtain the patient's written consent to contact their treating clinician to determine the appropriateness of study participation. We will not influence the decision patients make with their prescribing physician. All pharmacotherapy recommendations will be made in consultation with Dr. Murphy.
4. (a) Current clinically significant suicidality or (b) individuals who have engaged in suicidal behaviors within 6 months will be excluded and referred for appropriate clinical intervention.
5. Lifetime DSM-IV bipolar, schizophrenia or schizoaffective disorders; or Substance abuse in past 6 months.
6. Unwillingness of parents to make the commitment to accompany their child for multiple study visits.
7. Presence of a significant and/or unstable medical illness which might lead to hospitalization during the study.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2011-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Center for Neuropsychiatry, St. Petersburg, Florida, United States

REFERENCES:
- [Derived] Elliott SJ, Marshall D, Morley K, Uphoff E, Kumar M, Meader N. Behavioural and cognitive behavioural therapy for obsessive compulsive disorder (OCD) in individuals with autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2021 Sep 3;9(9):CD013173. doi: 10.1002/14651858.CD013173.pub2. PMID 34693989
- [Derived] Storch EA, Lewin AB, Collier AB, Arnold E, De Nadai AS, Dane BF, Nadeau JM, Mutch PJ, Murphy TK. A randomized controlled trial of cognitive-behavioral therapy versus treatment as usual for adolescents with autism spectrum disorders and comorbid anxiety. Depress Anxiety. 2015 Mar;32(3):174-81. doi: 10.1002/da.22332. Epub 2014 Nov 25. PMID 25424398

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cognitive Behavioral Therapy Condition | Treatment as Usual
Started | 16 | 15
Completed | 16 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavioral Therapy Condition | Treatment as Usual | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 15 | 31
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.75 (1.24) | 12.73 (1.49) | 12.74 (1.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 12 | 13 | 25
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 12 | 14 | 26
  Pacific Islander | 1 | 0 | 1
  Hispanic | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 16 | 15 | 31

OUTCOME MEASURES:

1. Primary Outcome: Pediatric Anxiety Rating Scale
Description: Scale range - 0 (minimum) to 25 (maximum). Higher scores represent worse anxiety symptom severity.
Time Frame: After an average of 16 weeks (Post-treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavioral Therapy Condition | Treatment as Usual
Number analyzed (Participants) | 16 | 15
units on a scale | 10.94 (3.91) | 13.93 (3.56)

2. Secondary Outcome: Anxiety Disorders Interview Schedule Clinical Severity Rating
Description: Scale range - 0 (minimum) to 8 (maximum). Higher scores represent worse anxiety symptom severity.
Time Frame: After an average of 16 weeks (Post-treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavioral Therapy Condition | Treatment as Usual
Number analyzed (Participants) | 16 | 15
units on a scale | 3.69 (1.35) | 5.33 (.9)

3. Secondary Outcome: Clinical Global Impression - Severity Scale
Description: Scale range - 0 (minimum) to 6 (maximum). Higher scores represent worse anxiety symptom severity.
Time Frame: After an average of 16 weeks (Post-treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavioral Therapy Condition | Treatment as Usual
Number analyzed (Participants) | 16 | 15
units on a scale | 2.88 (.72) | 3.67 (.82)

ADVERSE EVENTS:
Arm/Group | Cognitive Behavioral Therapy Condition | Treatment as Usual
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 0/16 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes